CLINICAL TRIAL: NCT06065085
Title: The Effect of Education Given to Individuals With Hypertension by Mobile Phone on DASH Diet Compliance, Quality of Life, Mindfulness and Stress
Brief Title: The Effect of Education Given to Individuals With Hypertension by Mobile Phone
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Trakya University (Other)
Responsible Party: Principal Investigator, Gulcan Meshur, PhD. Registered Nurse, Trakya University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2021/128
Record Dates: First submitted 2023-09-18; First posted 2023-10-03 (Actual); Last update posted 2023-10-03 (Actual); Status verified 2023-09

CONDITIONS: Hypertension; Mobile Education
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Mobile Education (Experimental): An education application was installed on the mobile phones of the experimental group. Individuals with hypertension were provided with a training for three months through the mobile application. Data collection forms were filled in by the individuals with hypertension in the experimental and controlled groups at the beginning and at the 3rd month via the mobile application.
  Interventions: Other: mobile education

INTERVENTIONS:
Other: mobile education — The study was conducted as a randomized controlled trial with 134 individuals with hypertension (68 experimental, 66 controlled) who applied a university hospital. The data were collected by "Patient Information Form", "Healthy Lifestyle Behaviour Scale II", "EQ-5D General Quality of Life Scale", "Mindful Attention Awareness Scale" and "Percieved Stress Scale" were used. An education application was installed on the mobile phones of the experimental group. Individuals with hypertension were provided with a training for three months through the mobile application. Data collection forms were filled in by the individuals with hypertension in the experimental and controlled groups at the beginning and at the 3rd month via the mobile application.

SUMMARY:
This study was planned as randomized controlled trial in order to evaluate the effect of the mobile education given to the individuals with hypertension on DASH diet compliance, healthy lifestyle behaviours, quality of life, mindfulness and stress levels.

The study was conducted as a randomized controlled trial with 134 individuals with hypertension (68 experimental, 66 controlled) who applied a university hospital in Edirne between the dates on 20.01.2022 and 18.05.2023. The data were collected by "Patient Information Form", "Healthy Lifestyle Behaviour Scale II", "EQ-5D General Quality of Life Scale", "Mindful Attention Awareness Scale" and "Percieved Stress Scale" were used. An education application was installed on the mobile phones of the experimental group. Individuals with hypertension were provided with a training for three months through the mobile application. Data collection forms were filled in by the individuals with hypertension in the experimental and controlled groups at the beginning and at the 3rd month via the mobile application. The data were analyzed in SPSS 26 (Statistical Package for the Social Sciences) program with the Shapiro-Wilk test, Student's t-test, Paired-Sample t-test, Chi-Square test, Fisher's Exact test, Fisher-Freeman-Halton test and Pearson correlation coefficient. The results were evaluated at % 95 confidence interval and the significance was evaluated at p<0,05 level.

ELIGIBILITY:
Inclusion Criteria:

* Those diagnosed with Primary Hypertension (at least 1 month ago),
* Over 18 years,
* No communication barriers,
* Being literate,
* Volunteering to participate in the research,
* Individuals with hypertension who own a smartphone.

Exclusion Criteria:

* under 18 years old,
* Having a communication barrier,
* Those with chronic kidney disease,
* Individuals with hypertension and heart failure.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 134 (Actual)
Dates: Start 2022-01-20 (Actual); Primary Completion 2023-05-18 (Actual); Study Completion 2023-08-10 (Actual)

PRIMARY OUTCOMES:
Mobile Education | three months
  The education given to individuals with hypertension via mobile phone was evaluated with healthy lifestyle behaviors, quality of life, stress and awareness scales.

SECONDARY OUTCOMES:
Healty Lifestyle Behaviour | three months
  The education given to individuals with hypertension via mobile phone was evaluated with the healthy lifestyle behaviors scale II.

OTHER OUTCOMES:
Quality of Life (EQ-5D General Quality of Life Scale) | three months
  The education given to individuals with hypertension via mobile phone was evaluated with EQ-5D General Quality of Life Scale.
Stress | three months
  The education given to individuals with hypertension via mobile phone was evaluated with Percieved Stress Scale .
Mindfulness | three months
  The education given to individuals with hypertension via mobile phone was evaluated with Mindful Attention Awareness Scale.

CONTACTS AND LOCATIONS:
Locations (1):
- Trakya Üniversitesi, Edirne, Merkez, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
It will be shared with the participants after it becomes published.